CLINICAL TRIAL: NCT05860933
Title: A Phase 1 Study to Evaluate the Effects of Multiple Doses of Itraconazole or Carbamazepine on the Single-Dose Pharmacokinetics of LY3537982 in Healthy Adult Subjects
Brief Title: A Study of the Effects of Itraconazole or Carbamazepine on LY3537982 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LOXO-RAS-22002; J3M-OX-JZQD (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-05-08; First posted 2023-05-16 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Healthy
MeSH Terms: interventions — Itraconazole; Carbamazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3537982 + Itraconazole (Part 1) (Experimental): LY3537982 administered orally alone followed by LY3537982 administered in combination with itraconazole orally.
  Interventions: Drug: LY3537982; Drug: Itraconazole
- LY3537982 + Carbamazepine (Part 2) (Experimental): LY3537982 administered orally alone followed by LY3537982 administered in combination with carbamazepine orally.
  Interventions: Drug: LY3537982; Drug: Carbamazepine

INTERVENTIONS:
Drug: LY3537982 — Administered orally.
  Other Names: Olomorasib
Drug: Itraconazole — Administered orally.
  Arms: LY3537982 + Itraconazole (Part 1)
Drug: Carbamazepine — Administered orally.
  Arms: LY3537982 + Carbamazepine (Part 2)

SUMMARY:
The main purpose of this study is to evaluate the effect of itraconazole and carbamazepine on LY3537982 when administered as multiple doses by conducting the blood tests to measure how much LY3537982 is in the bloodstream and how the body handles and eliminates LY3537982 in adult healthy participants. The study will also evaluate the safety and tolerability of LY3537982. The study is conducted in two parts. Participants will stay in the research center during the study, which will last about 11 and 15 days for part 1 and part 2, respectively, not including screening.

ELIGIBILITY:
Inclusion Criteria:

* Healthy status as defined by the absence of evidence of any clinically significant active or chronic disease
* Body mass index (BMI): 18.0 to 32.0 kilograms per square meter (kg/m²), inclusive

Exclusion Criteria:

* Females who are lactating or of childbearing potential
* Clinically significant history of any drug sensitivity, drug allergy, or food allergy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of LY3537982 administered with or without itraconazole | Predose on day 1 up to 72 hours postdose on day 9
  PK: Cmax of LY3537982 administered with or without itraconazole
PK: Area Under the Concentration-Time Curve (AUC) from Time 0 to Infinity (AUC[0-inf]) of LY3537982 administered with or without itraconazole | Predose on day 1 up to 72 hours postdose on day 9
  PK: AUC[0-inf] of LY3537982 administered with or without itraconazole
PK: AUC from Time 0 to time of the last measurable concentration (AUClast) of LY3537982 administered with or without itraconazole | Predose on day 1 up to 72 hours postdose on day 9
  PK: AUClast of LY3537982 administered with or without itraconazole
PK: Cmax of LY3537982 administered with or without carbamazepine | Predose on day 1 up to 72 hours postdose on day 13
  PK: Cmax of LY3537982 administered with or without carbamazepine
PK: AUC[0-inf] of LY3537982 administered with or without carbamazepine | Predose on day 1 up to 72 hours postdose on day 13
  PK: AUC[0-inf] of LY3537982 administered with or without carbamazepine
PK: AUClast of LY3537982 administered with or without carbamazepine | Predose on day 1 up to 72 hours postdose on day 13
  PK: AUClast of LY3537982 administered with or without carbamazepine

CONTACTS AND LOCATIONS:
Overall Officials: Yingying Guo-Avrutin, MD, PhD, Study Director — Loxo Oncology, Inc.
Locations (2):
- United States (2):
  - ICON Early Development Services, San Antonio, Texas
  - ICON Early Development Services, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No